CLINICAL TRIAL: NCT07107971
Title: Drug-Eluting Balloon Treatment Versus Guideline-Directed Medical Therapy for the Treatment of Lipid-Rich Plaques: A Randomized Controlled Trial
Brief Title: Drug-Eluting Balloon Treatment vs. Guideline-Directed Medical Therapy for the Treatment of Lipid-Rich Plaques
Acronym: DELETE-LRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Bimmer Claessen, Interventional Cardiologist, Department of Cardiology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL-009200
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Atheroscleroses; Cardiovascular Disease; Vulnerable Coronary Plaques; Vulnerable Plaque; Lipid-Rich Atherosclerosis of Coronary Artery; Acute Coronary Syndromes (ACS)
Keywords: Lipid-rich plaque; Vulnerable plaque; Near-infrared spectroscopy; Drug-coated balloon; Drug-eluting balloon; Paclitaxel-eluting balloon; Intravascular Ultrasound; Coronary computed tomography angiography; AI-QCT
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Cardiovascular Diseases; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: A total of 400 patients with acute coronary syndrome will be enrolled and undergo NIRS-IVUS imaging. Based on prior studies, approximately 50% are expected to have lipid-rich plaques (defined as maxLCBI4mm ≥325). These 200 patients will be randomized 1:1 to receive either drug-coated balloon treatment plus guideline-directed medical therapy or guideline-directed medical therapy alone. The remaining patients without lipid-rich plaques will be followed in an observational cohort within the DELETE-LRP study for long-term clinical outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Drug-coated balloon treatment of non-culprit lipid-rich plaque on top of guideline-directed medical therapy
  Interventions: Device: Paclitaxel-eluting balloon
- Control group (No Intervention): Guideline-directed medical therapy alone

INTERVENTIONS:
Device: Paclitaxel-eluting balloon — Participants in the intervention group will receive local treatment of non-obstructive, lipid-rich coronary plaques using a paclitaxel-coated drug-eluting balloon (DCB) in addition to guideline-directed medical therapy (GDMT). The DCB will be applied to plaques identified as high-risk based on near-infrared spectroscopy intravascular ultrasound (NIRS-IVUS) imaging, defined by a maxLCBI4mm ≥325. The balloon catheter diameter will be sized 1:1 according to the true lumen diameter as derived from IVUS. Balloon length will be sized to the LRP length as measured with IVUS including a 5 mm margin on each side. The balloon will be inflated at nominal pressure (6-8 ATM) during a period of at least 60 seconds, but preferably for 90 seconds if tolerated. A 5 mm margin is taken into account to differentiate between single or multiple LRPs within the same coronary artery.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to find out whether treating vulnerable plaques in the coronary arteries with a drug-coated balloon can make them less dangerous than using standard medication alone. The study includes adults with acute coronary syndrome (a type of heart problem caused by reduced blood flow in the coronary arteries).

The main questions the study aims to answer are:

* Does the drug-coated balloon reduce the amount of fat inside the plaque more than medication alone?
* Is this treatment safe for patients?

Participants will:

* Undergo imaging of their coronary arteries during their planned heart procedure (PCI)
* Be randomly assigned to receive either a drug-coated balloon treatment or no extra treatment
* Undergo a heart scan (CT scan of the coronary arteries) within 2 weeks and again around 9 months after the procedure.
* Undergo a second heart catherization 9 months later to examine changes in the plaque.

DETAILED DESCRIPTION:
Rationale:

Acute coronary syndromes (ACS) are often caused by rupture or erosion of certain high-risk vulnerable plaques. These plaques demonstrate specific features, such as a large lipid-rich necrotic core, a thin fibrous cap, and inflammation. Half of patients presenting with non-ST-segment elevation ACS have an additional vulnerable plaque, which increases their risk for non-culprit events during follow-up. Coronary intravascular ultrasound (IVUS) with the addition of near-infrared spectroscopy (NIRS) enables the identification of coronary lesions with high lipid content, quantified using the lipid-core burden index (LCBI) and is therefore able to distinguish plaques at risk to cause future non-culprit events. In addition, computed tomography coronary angiography (CCTA) is a non-invasive imaging modality that can identify high-risk plaque characteristics such as positive remodeling, low attentuation plaque, napkin-ring sign, and spotty calcification. Incorporating CCTA into this trial offers a unique opportunity to explore the potential of AI-based quantitative CT (AI-QCT) paramters by comparing them to IVUS-NIRS findings and clinical outcomes, which may support the future role of CCTA as a non-invasive tool for identifying and monitoring vulnerable plaques.

The main question remains whether local and systemic treatment of such high-risk plaques decreases the risk for adverse clinical outcome.

In our previous pilot study, DEBuT-LRP, we demonstrated that it was safe and feasible to treat vulnerable lipid-rich plaques with a drug-coated balloon (DCB) and that it was able to reduce the maximum LCBI on a 4 mm segment (maxLCBI4mm) after 9 months. In this randomized controlled trial, we intend to investigate the impact of DCB treatment on the maxLCBI4mm of lipid-rich plaques when compared to guideline-directed medical therapy alone.

Objective:

To test the hypothesis that paclitaxel-coated balloon treatment of non-obstructive non-culprit vulnerable lipid-rich plaques (LRP) leads to a greater reduction of the lipid-core burden index than guideline-directed medical therapy alone.

Study design:

A prospective two-arm randomized controlled trial.

Study population:

Patients older than 18 years with ACS who are scheduled for invasive percutaneous coronary intervention (PCI) of a native coronary artery.

Intervention:

DCB treatment of LRP in addition to guideline-directed medical therapy (GDMT).

Main study parameters:

The main study endpoint is the difference in maxLCBI4mm reduction from baseline to 9 months follow-up compared between the two randomization groups.

Secondary study endpoints are clinical safety endpoints (1. Flow-limiting dissection related to DCB-treatment necessitating bail-out stenting; 2. Periprocedural myocardial infarction; 3. Bleeding; 4. LRP lesion failure: cardiovascular death, myocardial infarction or repeat revascularization related to the index LRP, 5. Patient-oriented outcome: all-cause death, myocardial infarction or repeat revascularization) and imaging endpoints (1. IVUS-derived parameters; 2. QCA endpoints; 3. NIRS analyses of non-treated vessels; 4. CCTA-derived parameters).

ELIGIBILITY:
Inclusion Criteria:

* Presenting with acute coronary syndrome (ACS);
* Successful PCI of a native coronary artery or major side branch;
* At least 2 native coronary arteries are accessible for invasive coronary imaging; i.e. not totally occluded and >2 mm and <6 mm reference vessel diameter.

Exclusion Criteria:

* Hemodynamically unstable (presence of cardiogenic shock, need for intubation, need for inotropes);
* Known hypersensitivity to paclitaxel;
* Procedural complications of the index PCI;
* Known renal insufficiency, i.e. eGFR <30 mL/min/1.73 m2;
* Hypersensitivity or allergy to contrast with inability to administer steroid and antihistamine premedication;
* Presence of a comorbid condition with a life expectancy of less than one year;
* Body weight >250 kg;
* Subject belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff) or is unable to read or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Difference in maxLCBI4mm of the target LRP | From baseline to 9 month follow-up.
  The mean difference in maxLCBI4mm of the target LRP between baseline and 9 month follow-up compared between the two randomization groups.

SECONDARY OUTCOMES:
Difference in maxLCBI4mm in non-treated LRPs | From baseline to 9 month follow-up.
  The change in maxLCBI4mm as measured with IVUS/NIRS from baseline to 9 month follow-up in identified additional LRPs that are not treated with DCB.
The change in IVUS- and angiography-derived measurements | From baseline to 9 month follow-up.
  The change in IVUS- and angiography-derived measurements (plaque burden, minimal lumen area, mean plaque area, diameter stenosis and minimal lumen diameter) between baseline and 9 month follow-up.
The change in CCTA-derived measurements | From baseline to 9 month follow-up.
  The change in CCTA-derived measurements using AI-QCT (total plaque volume, noncalcified plaque volume, calcified plaque volume, lumen volume and presence of the following high-risk plaque features: positive remodeling [remodeling index >1.1] and low-density plaque).
Flow-limiting dissection necessitating bail-out stent implantation | From baseline to 9 month follow-up.
  Flow-limiting dissection necessitating bail-out stent implantation.
Periprocedural myocardial infarction | From baseline to 9 month follow-up.
  Procedure-related myocardial infarction is defined according to the Fourth Universal Definition for Myocardial Infarction. Periprocedural myocardial infarction has occurred when an elevation of cTn values > 5 times of the 99th percentile URL in patients with normal baseline values is measured within a time window up to 48 hours post-procedure.
  Patients with elevated pre-procedural cTn values, in whom the pre-procedural cTn level are stable (≤ 20% variation) or falling, must meet the criteria for a >5 or >10 fold increase and manifest a change from the baseline value of >20%. In addition with at least one of the following:
  * New ischaemic ECG changes;
  * Development of new pathological Q waves;
  * Imaging evidence of loss of viable myocardium that is presumed to be new and in a pattern consistent with an ischaemic aetiology;
  * Angiographic findings consistent with a procedural flow-limiting complication.
Bleeding (BARC-3 and -5) | From baseline to 5 year follow-up.
  The occurence of BARC Type 3 or 5 bleeding events.
LRP lesion failure | From baseline to 5 year follow-up.
  LRP lesion failure, defined as the occurence of cardiovascular death, myocardial infarction, or ischemia-driven revascularization related to an identified non-culprit LRP lesion.
Patient-oriented composite outcome | From baseline to 5 year follow-up.
  Patient-oriented composite outcome, defined as the occurrence of all-cause mortality, myocardial infarction, or any repeat revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Bimmer E.P.M. Claessen, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands